CLINICAL TRIAL: NCT03864367
Title: Mobile Weight-Support Therapy (MWeST) for Mobility After Geriatric Fracture
Acronym: MWeST
Status: Withdrawn | Type: Observational
Why Stopped: PI decided to end the study
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201805050
Record Dates: First submitted 2019-01-31; First posted 2019-03-06 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Distal Femur Fracture
MeSH Terms: conditions — Femoral Fractures, Distal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Device: This group will use the MWeST lift device along with regular physical therapy. The lift device is the Prism Medical FGA-700 Bariatric Floor Lift including a sling to assist in walking.
  Interventions: Device: Device - Prism Medical FGA-700 Bariatric Floor Lift
- Control: This group will only receive regular physical therapy.

INTERVENTIONS:
Device: Device - Prism Medical FGA-700 Bariatric Floor Lift — This group will be using a Mobile Weight-Support Therapy (MWeST) device (the Prism Medical FGA-700 Bariatric Floor Lift) to determine if it improves mobilization of older patients with traumas of their legs.
  Groups: Device

SUMMARY:
This is a two-year study proposal to assess feasibility of MWeST (Mobile Weight-Support Therapy) implementation after geriatric fracture and its effects on functional and patient-reported outcomes.

The goal of this study is to improve mobilization of geriatric lower extremity trauma patients, with the aim of improving overall functional and patient-reported outcomes while decreasing complications and readmissions. Almost 50% of the adult population in the United States has osteopenia or osteoporosis, with over 2 million fragility fractures per year and a projected $25 billion in costs by 2025. These patients are at high risk for readmission due to complications, and at increased risk of mortality with these complications. Sarcopenia, a generalized loss of skeletal muscle associated with aging, has also been associated with increased disability and increased risk of future fracture in these patients. The investigator's study aims to assess the value of weight-support therapy for geriatric patients with lower extremity trauma in improving their overall risk of future injury and disability.

DETAILED DESCRIPTION:
The goal of this study is to improve mobilization of geriatric lower extremity trauma patients, with the aim of improving overall functional and patient-reported outcomes while decreasing complications and readmissions. Almost 50% of the adult population in the United States has osteopenia or osteoporosis, with over 2 million fragility fractures per year and a projected $25 billion in costs by 2025. These patients are at high risk for readmission due to complications, and at increased risk of mortality with these complications. Sarcopenia, a generalized loss of skeletal muscle associated with aging, has also been associated with increased disability and increased risk of future fracture in these patients. The investigator's study aims to assess the value of weight-support therapy for geriatric patients with lower extremity trauma in improving their overall risk of future injury and disability.

ELIGIBILITY:
Inclusion Criteria:

* 55 and older
* distal femur fracture
* able to walk prior to fracture

Exclusion Criteria:

* patients unable to walk without any assistive devices post-injury
* patients too medically unstable to participate in physical therapy

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is anyone 55 years of age and older with a distal femur fracture.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
Walking with device | 1 year
  Determining if the Mobile Weight-Support device helps improve mobility after injury compared to walking without device.

CONTACTS AND LOCATIONS:
Overall Officials: ANNA N MILLER, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
This is a single site study.